CLINICAL TRIAL: NCT00345774
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Short-Term Efficacy and Safety of PRX-08066 in Patients With Pulmonary Hypertension and Chronic Obstructive Pulmonary Disease
Brief Title: Safety and Effectiveness of PRX-08066 in Patients With Pulmonary Hypertension and Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Epix Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRX-CP-017
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Pulmonary Hypertension; Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary Hypertension; PH; Pulmonary Arterial Hypertension; PAH; Chronic Obstructive Pulmonary Disease; COPD; PRX-08066; Predix
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive; Pulmonary Arterial Hypertension | interventions — 5-((4-(6-chlorothieno(2,3-d)pyrimidin-4-ylamino)piperidin-1-yl)methyl)-2-fluorobenzonitrile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PRX-08066

SUMMARY:
This study is being conducted to see if PRX-08066 can lower pulmonary artery pressures in patients with pulmonary hypertension associated with chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

1. 25 to 79 years old.
2. Provide voluntary written informed consent to participate.
3. Smoking history of at least 10 pack years (1 pack of cigarettes per day for 10 years).
4. Diagnosis of chronic obstructive pulmonary disease.
5. Become short of breath with physical activity.
6. Elevated systolic pulmonary artery pressures.
7. Not pregnant, nursing, or planning a pregnancy.

Exclusion Criteria:

1. Left ventricular ejection fraction <30%.
2. Heart attack or stroke within the last 6 months.
3. History of lung resection surgery.
4. Use of supplemental oxygen >20 hours/day.
5. Blood donation or significant blood loss within the last 56 days.
6. Plasma donation within the last 14 days.
7. Use of any drugs for another research study within the last 30 days.
8. Use of vasodilators, long acting nitrates, prostacyclin analogs, endothelin antagonists, or phosphodiesterase inhibitor drugs within the last 14 days.
9. Positive blood screen Hepatitis B surface antigen (HBsAg) or Hepatitis C Antibody.
10. Major surgery within the last 28 days.
11. Any other medical condition that may jeopardize the safety of the subject, the validity of the study results, or interfere with the completion of the study according to the protocol.

Ages: 25 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2006-06; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Systolic Pulmonary Artery Pressure

SECONDARY OUTCOMES:
Safety
6 minute walk distance
Borg Dyspnea Index
BDI/TDI
Echocardiograms
Spirometry
Oxygen saturation
WHO functional classification

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Arizona Pulmonary Specialists, Ltd., Phoenix, Arizona
  - University of California-Davis Medical Group, Sacramento, California
  - University Clinical Research-DeLand, LLC, DeLand, Florida
  - Central Medical Group, PA, Tamarac, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Atlanta Insitute for Medical Research, Decatur, Georgia
  - Pulmonary Consultants of North Idaho, Coeur d'Alene, Idaho
  - Loyola University Medical Center Foster McGraw Hospital, Maywood, Illinois
  - Veritas Clinical Specialities, Topeka, Kansas
  - Tufts New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Pulmonary Critical Care Unit, Boston, Massachusetts
  - Buffalo Cardiology and Pulmonary Associates, P.C., Williamsville, New York
  - American Health Research, Charlotte, North Carolina
  - South Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Morgantown Pulmonary Clinical Research, Morgantown, West Virginia
  - Heart Care Associates, LLC, Milwaukee, Wisconsin